CLINICAL TRIAL: NCT04415359
Title: Evaluation of the Evolution of Pregnancies in the First Trimester Following a Medically Assisted Procreation (MAR) Management During a COVD-19 Pandemic Period
Brief Title: Evaluation of the Evolution of Pregnancies in the First Trimester Following MAR Management During a COVD-19 Pandemic Period
Acronym: AMPCOVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7789
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-05

CONDITIONS: Covid-19
Keywords: COVID-19; SARS-CoV-2; ARDS; ICU; Pregnant women; Pregnancy; Fetus; Middle East Respiratory Syndrome; MERS; Maternal respiratory impairment; Medical Assisted Procreation; MAR; Frozen embryos
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Because of the physiological changes inherent in pregnancy, pregnant women with lower respiratory tract infections often have more worrisome outcomes compared to non-pregnant individuals, including a higher rate of hospital and intensive care unit admissions.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in a Medically Assisted Procreation (MAR) protocol aged between 18 and 43 years of age
* Patient who has already signed a consent to management

Exclusion Criteria:

* Patient who expressed opposition to participating in the study

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: Patient included in MAR protocol aged between 18 and 43 years of age who has already signed a consent to management
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Study of the evolution of pregnancies in the first trimester following MAR management during a COVD-19 pandemic period | 12th week of Amenorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Service Clinico biologique d'Assistance Médicale à La Procréation, Strasbourg, France